CLINICAL TRIAL: NCT02382419
Title: Expanded Phase II Trial of a Carrageenan-Containing Gel for Prevention of HPV Infection
Brief Title: Carrageenan-Containing Gel in Reducing the Rate of HPV Infection in Healthy Participants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator Decided to stop recruitment in the trial.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark H. Einstein, MD, MS, FACS, FACOS, Professor and Chair Department of Obstetrics, Gynecology and Women's Health, Assistant Dean, Clinical Research Unit, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20150002694; NCI-2015-00209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20150002694 (Other: Rutgers New Jersey Medical School); R01CA148966 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2015-02-26; First posted 2015-03-06 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Healthy Subject; Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (carrageenan-containing gel) (Experimental): Participants apply carrageenan-containing gel vaginally within 12 hours prior to each vaginal sex act and as soon as possible within 12 hours after each vaginal sex act and use condoms for 12 months.
  Interventions: Drug: carrageenan-containing gel; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm II (placebo gel) (Placebo Comparator): Participants apply placebo gel vaginally within 12 hours prior to each vaginal sex act and as soon as possible within 12 hours after each vaginal sex act and use condoms for 12 months.
  Interventions: Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: carrageenan-containing gel — Applied vaginally
  Other Names: Divine 9 with Carragel
  Arms: Arm I (carrageenan-containing gel)
Other: Placebo — Applied vaginally
  Other Names: PLCB
  Arms: Arm II (placebo gel)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well carrageenan-containing gel (vaginal gel) works in reducing the rate of human papilloma virus (HPV) infection in healthy participants. Carrageenans, which are naturally derived from seaweed, are enhancements to natural lubrication and may be effective in blocking HPV infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the overall efficacy of the intervention in reducing the rate of incident cervical HPV infection.

SECONDARY OBJECTIVES:

I. Perform in vitro exploratory testing of how long after vaginal application the drug retains biological activity by collecting cervicovaginal lavage (CVL) at different times and spiking the samples with HPV pseudovirions (PsVs) and measuring PsV entry into target cells.

II. These studies will be expanded to test multiple HPV types and to examine whether the anti-HPV activity of the intervention is preserved in the setting of semen.

III. Store swabs to potentially test candidate biomarkers of microbicide efficacy and safety.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants apply carrageenan-containing gel vaginally within 12 hours prior to each vaginal sex act and as soon as possible within 12 hours after each vaginal sex act and use condoms for 12 months.

ARM II: Participants apply placebo gel vaginally within 12 hours prior to each vaginal sex act and as soon as possible within 12 hours after each vaginal sex act and use condoms for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women of all ethnicities and races with an intact cervix are eligible for this trial
* Engaging in three or more intercourse events (defined as having penile-vaginal intercourse) per month; subjects must consent not to douche or use any vaginal products, including tampons, for 24 hours before enrollment and study visits
* Normal Pap or Atypical Squamous Cells of Undetermined Significance (ASCUS) Pap test with HPV deoxyribonucleic acid (DNA) negative by reflex testing via Hybrid Capture 2 (Digene Corp., Gaithersburg, MD), a standard clinical assay within clinically acceptable screening guidelines (American Cancer Society [ACS]/American Society for Colposcopy and Cervical Pathology [ASCCP] 2012 Screening Guidelines)
* Using an adequate method of contraception for at least 3 months with no changes and will remain on the contraception for the duration of the trial; an adequate method of contraception is defined as either a hormonal based method (except vaginal rings); an intrauterine device (IUD) (inserted at least 30 days prior to enrollment); female sterilization; or sexual activity with a partner who had a vasectomy
* Speaks either English or Spanish, living in or near Newark with no plans to move in the next year, able to sign consent and complete questionnaires with aid of trained personnel

Exclusion Criteria:

* Prior use of an HPV vaccine

  * Women in the vaccine-eligible age range cannot have received vaccine prior to enrollment, but will be offered HPV vaccination at the end of the study; in brief, we are interested in the efficacy of intervention in preventing HPV in the absence of HPV vaccination, since most women worldwide who might utilize intervention will not have been vaccinated; this includes United States (US) women in the vaccine "catch-up" 19-26 year old age group (beyond the age groups eligible for Vaccines for Children- funded vaccination) who have so far had very low (< 10%) vaccine uptake; it also includes the entire group of US women > 26 years of age; moreover, it includes women of all ages in developing countries, who most need an HPV prevention strategy, but may never be vaccinated; it should be noted that delaying vaccination in women 19-26 years of age by one year is safe and reasonable, since there is insufficient data to establish a recommendation for or against universal vaccination in this age group as concluded by an American Cancer Society expert panel, which includes the Principal Investigator (PI) of this protocol, Dr. Mark Einstein; it is anticipated that if the intervention gel is efficacious, HPV vaccinated women would need to be studied in a similar future trial with power analysis taking into account vaccine effectiveness as well
* Any previous surgical excision of cervical intraepithelial neoplasia (CIN) or hysterectomy
* A serious, concomitant disorder, including active systemic infection requiring treatment
* Prior history of or current malignancy other than adequately treated skin cancer (squamous cell cancer or basal cell carcinoma)
* Documented or suspected immunosuppressive disorder or autoimmune disease
* Any significant cardiac, hepatic or renal disease
* Pregnant and/or breast-feeding
* Recent (within 4 weeks of screening) or concomitant long term treatment with systemic steroids, immunosuppressive/immunomodulating drugs (e.g. cyclosporine, corticosteroids)

  * Intranasal, inhaled and/or topical steroids are permissible
* Documented human immunodeficiency virus (HIV) infection, genital warts, chancroid, or pelvic inflammatory disease that will require long term treatment
* Active genital ulcers
* Use of an investigational drug in the 3 months prior to screening and must agree to not participate in any drug or device study while enrolled in this study
* Any known allergy or hypersensitivity to vaginal lubricants or any component of study product

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Rate of incident cervical HPV infection | Up to 1 year
  The primary analysis will be based upon the intent to treat approach. The cumulative incidence of HPV infection for each treatment group will be estimated as described above and the percent reduction in incidence due to intervention will be computed along with the corresponding one-sided 80% lower confidence bound.

SECONDARY OUTCOMES:
Cumulative incidence rates of HPV in the target population (using data from the placebo group) | At 1 year
  Multivariate logistic regression models that incorporate additional subject data (e.g., frequency of intercourse and number of recent sex partners, anal sex, and smoking behavior) will be fit to the data to control for potential imbalances in subject characteristics that may occur despite randomization with HPV infection status as the binary dependent variable. A generalized estimating equation approach will also be used to model treatment effect on infection with multiple HPV types.
Subject adherence as measured by monthly applicator collection and counting | Up to 1 year
  Will perform a per protocol analysis including only "adherent" subjects, defined as subjects who report gel use as recommended (within one hour of intercourse) in > 50% of all vaginal intercourse acts. Will perform additional analyses to identify any imbalances in subject characteristics across groups, and in secondary analyses using logistic regression models to incorporate this as above.
Behavioral characteristics assessed by questionnaires | Up to 1 year
  Multivariate logistic regression models that incorporate additional subject data (e.g., frequency of intercourse and number of recent sex partners, anal sex, and smoking behavior) will be fit to the data to control for potential imbalances in subject characteristics that may occur despite randomization with HPV infection status as the binary dependent variable. A generalized estimating equation approach will also be used to model treatment effect on infection with multiple HPV types.
Biological activity of carrageenan-containing gel or placebo as measured by CVL at different times and spiking the samples with HPV PsVs and measuring PsV entry into target cells | Baseline to up to 12 months
  Changes in this variable at each time point relative to baseline will be compared between groups using analysis of covariance models to adjust for baseline level. In addition, linear mixed effects models will be fit to all the repeated measurements to evaluate and compare trends over time while adjusting for the within-subject correlation in the data.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Einstein, Principal Investigator — Rutgers University
Locations (1):
- Rutgers New Jersey Medical School, Newark, New Jersey, United States